CLINICAL TRIAL: NCT01852019
Title: A Study of the Transition From IV Cangrelor to Oral Prasugrel, and Prasugrel to Cangrelor, in Patients With Coronary Artery Disease.
Brief Title: Cangrelor Prasugrel Transition Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: MDCO-CAN-13-01
Record Dates: First submitted 2013-05-06; First posted 2013-05-13 (Estimated); Results first posted 2015-05-28 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease | interventions — cangrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Day 1 - Cangrelor + Prasugrel (60mg) post infusion (Experimental): Cangrelor IV + Oral prasugrel (60mg) administered within 5 minutes after cangrelor IV discontinuation
  Interventions: Drug: Cangrelor; Drug: Prasugrel
- Day 8 - Prasugrel (10mg) Dosing (5 doses) (Experimental): Prasugrel discontinued 48h (n=6) prior to initiation of cangrelor infusion (2h)
  Interventions: Drug: Cangrelor; Drug: Prasugrel
- Day 1 - Cangrelor + Prasugrel (60mg) at 1.5h (Experimental): Cangrelor IV + oral prasugrel (60mg) administered at 1.5h after the cangrelor infusion start time.
  Interventions: Drug: Cangrelor; Drug: Prasugrel
- Day 1 - Cangrelor + Prasugrel (60mg) a 1.0h (Experimental): Cangrelor IV + oral prasugrel (60mg) administered at 1.0h after the cangrelor infusion start time.
  Interventions: Drug: Cangrelor; Drug: Prasugrel
- Day 8 - Prasugrel (10mg) Dosing (6 doses) (Experimental): Prasugrel discontinued 24h prior to initiation of cangrelor infusion (2h)
  Interventions: Drug: Cangrelor; Drug: Prasugrel

INTERVENTIONS:
Drug: Cangrelor — Cangrelor IV administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
Drug: Prasugrel — Day 1: Subjects received prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects will be given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.

SUMMARY:
To demonstrate that patients treated with cangrelor can be directly switched to oral prasugrel and that patients treated with prasugrel can be switched to cangrelor without a significant decrease in the extent of inhibition of platelet aggregation.

ELIGIBILITY:
Inclusion Criteria:

1. greater than / equal to 18 and less than 75 years of age
2. stable coronary artery disease defined by the following criteria

   1. Previous myocardial infarction defined by admission to the hospital with elevation of markers of injury or the presence of pathologic Q waves on at least 2 contiguous electrocardiogram (ECG) leads.

      OR
   2. Previous revascularization by percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG).

      AND
   3. Treatment with aspirin (ASA) 81 mg daily.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Schneider, Principal Investigator — University of Vermont Medical Center
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Day 1 - Cangrelor + Prasugrel (60mg) Post Infusion: Cangrelor IV + Oral prasugrel (60mg) administered within 5 minutes after cangrelor IV discontinuation
  cangrelor: Cangrelor IV is administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects will receive prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects will be given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
- Day 1 - Cangrelor + Prasugrel (60mg) a 1.0h: Cangrelor IV + oral prasugrel (60mg) administered at 1.0h after the cangrelor infusion start time.
  cangrelor: Cangrelor IV is administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects will receive prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects will be given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
- Day 1 - Cangrelor + Prasugrel (60mg) at 1.5h: Cangrelor IV + oral prasugrel (60mg) administered at 1.5h after the cangrelor infusion start time.
  cangrelor: Cangrelor IV is administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects will receive prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects will be given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
- Day 8 - Prasugrel (10mg) Dosing (5 Doses): Prasugrel discontinued 48h (n=6) prior to initiation of cangrelor infusion (2h)
  cangrelor: Cangrelor IV is administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects will receive prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects will be given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
- Day 8 - Prasugrel (10mg) Dosing (6 Doses): Prasugrel discontinued 24h prior to initiation of cangrelor infusion (2h)
  cangrelor: Cangrelor IV is administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects will receive prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects will be given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
Period: Day 1
Arm/Group | Day 1 - Cangrelor + Prasugrel (60mg) Post Infusion | Day 1 - Cangrelor + Prasugrel (60mg) a 1.0h | Day 1 - Cangrelor + Prasugrel (60mg) at 1.5h | Day 8 - Prasugrel (10mg) Dosing (5 Doses) | Day 8 - Prasugrel (10mg) Dosing (6 Doses)
Started | 3 | 3 | 6 | 0 | 0
Completed | 3 | 3 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Day 8
Arm/Group | Day 1 - Cangrelor + Prasugrel (60mg) Post Infusion | Day 1 - Cangrelor + Prasugrel (60mg) a 1.0h | Day 1 - Cangrelor + Prasugrel (60mg) at 1.5h | Day 8 - Prasugrel (10mg) Dosing (5 Doses) | Day 8 - Prasugrel (10mg) Dosing (6 Doses)
Started | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population
Groups:
- Day 8 - Prasugrel (10mg) Dosing (5 Doses): Prasugrel discontinued 48h prior to initiation of cangrelor infusion (2h)
  Cangrelor: Cangrelor IV is administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects will receive prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects will be given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
- Total: Total of all reporting groups
Arm/Group | Day 8 - Prasugrel (10mg) Dosing (6 Doses) | Day 8 - Prasugrel (10mg) Dosing (5 Doses) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (6.47) | 67.3 (4.37) | 64.8 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Extent of Preservation of Inhibitory Effect After Transition From Cangrelor to Prasugrel Compared With Effect Observed With Prasugrel Alone (Reference Timepoint)
Description: A reference point for the effect of prasugrel alone was chosen for comparison and designated the final draw on study Day 1 (3.5 or 4.0 hours after cangrelor had been discontinued) as the reference for the effect of prasugrel. The extent of aggregation in the presence or absence of the study drugs was examined for each of the endpoints using light transmittance aggregometry (LTA) and expressed as % aggregation in response to 20 micromolar (μM) adenosine diphosphate (ADP) at 300 seconds (final/terminal aggregation response).
Time Frame: Day 1 measures taken at timepoints after cangrelor infusion end to end of Day 1 measures.
Population: Subjects treated with cangrelor and prasugrel were used for the analysis and presentation of data.
Measure: Mean (Standard Deviation); unit: % aggregation
Groups:
- Day 1 - Cangrelor + Prasugrel (60mg) Post Infusion (2.0h): Cangrelor IV + Oral prasugrel (60mg) were administered within 5 minutes after cangrelor IV discontinuation
  cangrelor: Cangrelor IV was administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects received prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects were given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
- Day 1 - Cangrelor + Prasugrel (60mg) at 1.5h: Cangrelor IV + oral prasugrel (60mg) was administered at 1.5h after the cangrelor infusion start time.
  cangrelor: Cangrelor IV was administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects received prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects were given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
- Day 1 - Cangrelor + Prasugrel (60mg) a 1.0h: Cangrelor IV + oral prasugrel (60mg) were administered at 1.0h after the cangrelor infusion start time.
  cangrelor: Cangrelor IV was administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects received prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects were given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
Arm/Group | Day 1 - Cangrelor + Prasugrel (60mg) Post Infusion (2.0h) | Day 1 - Cangrelor + Prasugrel (60mg) at 1.5h | Day 1 - Cangrelor + Prasugrel (60mg) a 1.0h
Number analyzed (Participants) | 3 | 6 | 3
% aggregation
  Prasugrel Reference (6.0h or 5.5 h) | 1.0 (1.0) | 2.8 (3.1) | 5.0 (6.2)
  2.25 h | 27 (20) | 25 (15) | 45 (24)
  2.5 h | 56 (6.7) | 42 (27) | 62 (3.8)
  2.75 h | 64 (2.1) | 31 (33) | 69 (4.6)
  3.0 h | 58 (14) | 24 (26) | 51 (5.1)
  4.0 h | 1.0 (1.7) | 10 (15) | 15 (18)

2. Primary Outcome: Extent of Preservation of Inhibitory Effect of Cangrelor Treatment After Prasugrel, Compared to Treatment With Cangrelor Alone
Description: A reference point for the inhibitory effect of cangrelor alone was chosen for comparison and designated the first draw during the cangrelor infusion (1.0 or 1.5 hours) or within 5 minutes post cangrelor infusion on Day 1. The extent of aggregation was observed during the cangrelor infusion on Day 8, either 24 or 48 hours after discontinuation of prasugrel using light transmittance aggregometry (LTA) and expressed as % aggregation in response to 20 μM adenosine diphosphate (ADP) at 300 seconds (final/terminal aggregation response).
Time Frame: Day 8 - at 1.0 and 2.0 hours after initiation of cangrelor infusion
Population: Subjects treated with cangrelor and prasugrel were used for the analysis and presentation of data.
Measure: Mean (Standard Deviation); unit: % aggregation
Groups:
- Day 8 - Prasugrel (10mg) Dosing (6 Doses): Prasugrel was discontinued 24h prior to initiation of cangrelor infusion (2h)
  Cangrelor: Cangrelor IV was administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects received prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects were given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
- Day 8 - Prasugrel (10mg) Dosing (5 Doses): Prasugrel was discontinued 48h prior to initiation of cangrelor infusion (2h)
  Cangrelor: Cangrelor IV iwas administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects received prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects were given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
Arm/Group | Day 8 - Prasugrel (10mg) Dosing (6 Doses) | Day 8 - Prasugrel (10mg) Dosing (5 Doses)
Number analyzed (Participants) | 6 | 6
% aggregation
  1.0 h | 0.5 (0.8) | 1.3 (2.0)
  2.0 h | 0.0 (0.0) | 1.0 (1.4)

3. Secondary Outcome: Extent of Preservation of Inhibitory Effect After Transition From Cangrelor to Prasugrel Compared With Effect Observed With Prasugrel Alone (Reference Timepoint)
Description: A reference point for the effect of prasugrel alone was chosen for comparison and designated the final draw on study Day 1 (3.5 or 4.0 hours after cangrelor had been discontinued) as the reference for the effect of prasugrel. The extent of aggregation in the presence of absence of the study drugs was examined for each of the endpoints as assessed by platelet reaction units (PRU) from the VerifyNow P2Y12 assay.
Time Frame: Day 1 measures taken at timepoints after cangrelor infusion end to end of Day 1 measures.
Population: Subjects treated with cangrelor and prasugrel were used for the analysis and presentation of data.
Measure: Mean (Standard Deviation); unit: platelet reaction units (PRU)
Arm/Group | Day 1 - Cangrelor + Prasugrel (60mg) Post Infusion (2.0h) | Day 1 - Cangrelor + Prasugrel (60mg) at 1.5h | Day 1 - Cangrelor + Prasugrel (60mg) a 1.0h
Number analyzed (Participants) | 3 | 6 | 3
platelet reaction units (PRU)
  Prasugrel Reference (6.0h or 5.5h) - PRU | 7.7 (12) | 41 (42) | 74 (60)
  2.25h - PRU | 91 (82) | 82 (39) | 151 (77)
  2.5h - PRU | 242 (50) | 181 (70) | 269 (38)
  2.75h - PRU | 267 (25) | 134 (94) | 285 (35)
  3.0h - PRU | 239 (50) | 127 (124) | 242 (32)
  4.0h - PRU | 20 (31) | 56 (68) | 117 (77)

4. Secondary Outcome: Extent of Preservation of Inhibitory Effect of Cangrelor Treatment After Prasugrel, Compared to Treatment With Cangrelor Alone
Description: A reference point for the inhibitory effect of cangrelor alone was chosen for comparison and designated the first draw during the cangrelor infusion (1.0 or 1.5 hours) or within 5 minutes post cangrelor infusion on Day 1. The extent of aggregation was observed during the cangrelor infusion on Day 8, either 24 or 48 hours after discontinuation of prasugrel as assessed by platelet reaction units (PRU) from the VerifyNow P2Y12 assay.
Time Frame: Day 8 - at 1.0 and 2.0 hours after initiation of cangrelor infusion
Population: Subjects treated with cangrelor and prasugrel were used for the analysis and presentation of data.
Measure: Mean (Standard Deviation); unit: platelet reaction units (PRU)
Arm/Group | Day 8 - Prasugrel (10mg) Dosing (6 Doses) | Day 8 - Prasugrel (10mg) Dosing (5 Doses)
Number analyzed (Participants) | 6 | 6
platelet reaction units (PRU)
  1.0 h - PRU | 6.3 (6.6) | 8.3 (5.4)
  2.0 h - PRU | 4.7 (2.6) | 13 (18)

5. Secondary Outcome: Bleeding Events in Accordance With the GUSTO Scale
Description: Bleeding was assessed by history, physical exam, and complete blood count (CBC) that was performed on study Days 1 and 8. Reports of bleeding were to be evaluated by performance of a CBC. Bleeding was to be reported as recommended and quantified in accordance with the GUSTO criteria [The GUSTO Investigators, 1993].
Time Frame: Day 1 through Day 8
Measure: Number; unit: participants
Groups:
- Day 8 - Prasugrel (10mg) Dosing (5 Doses): Prasugrel was discontinued 48h prior to initiation of cangrelor infusion (2h)
  Cangrelor: Cangrelor IV was administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects received prasugrel (60 mg) either during the initial cangrelor infusion (at 1.0 hours or 1.5 hours after infusion start) or within 5 minutes of discontinuing the cangrelor infusion.
  Subjects were given either 5 or 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
Arm/Group | Day 8 - Prasugrel (10mg) Dosing (6 Doses) | Day 8 - Prasugrel (10mg) Dosing (5 Doses)
Number analyzed (Participants) | 6 | 6
participants
  Mild | 1 | 0
  Moderate | 0 | 0
  Life-threatening/Severe | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening through Follow-up Period
Description: Follow-up period:
  Each subject was contacted by telephone 5 to 7 days after Study Day 8 to assess adverse event (AEs) / serious adverse events (SAEs) and to ensure that any previously identified AEs/SAEs had resolved.
Groups:
- Day 1 - Prasugrel (60mg) at 1.5 Hrs: Cangrelor: Cangrelor IV was administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects received prasugrel (60 mg) during the initial cangrelor infusion (at 1.5 hours after infusion start).
- Day 1 - Prasugrel (60mg) at 1.0 hr: Cangrelor: Cangrelor IV was administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects received prasugrel (60 mg) during the initial cangrelor infusion (at 1.0 hour after infusion start).
- Day 1 - Prasugrel (60mg) - Post Infusion (2.0 hr): Cangrelor: Cangrelor IV was administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
  Prasugrel: Day 1: Subjects received prasugrel (60 mg) post infusion, [at 2.0 hrs, (within 5 minutes of discontinuing the cangrelor infusion)].
- Day 8 - Prasugrel (10mg) Dosing (6 Doses): Prasugrel was discontinued 24h prior to initiation of cangrelor infusion (2h)
  Subjects were given 6 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
  Cangrelor: Cangrelor IV was administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
- Day 8 - Prasugrel (10mg) Dosing (5 Doses): Prasugrel was discontinued 48h prior to initiation of cangrelor infusion (2h)
  Subjects were given 5 additional 10-mg doses to be taken every 24 hours between Day 1 and Day 8.
  Cangrelor: Cangrelor IV was administered as a 30 µg/kg bolus, followed by 4 µg/kg/min infusion for two hours on study Days 1 and 8
Arm/Group | Day 1 - Prasugrel (60mg) at 1.5 Hrs | Day 1 - Prasugrel (60mg) at 1.0 hr | Day 1 - Prasugrel (60mg) - Post Infusion (2.0 hr) | Day 8 - Prasugrel (10mg) Dosing (6 Doses) | Day 8 - Prasugrel (10mg) Dosing (5 Doses)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/3 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 0/3 | 0/3 | 0/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Day 1 - Prasugrel (60mg) at 1.5 Hrs (N=6) | Day 1 - Prasugrel (60mg) at 1.0 hr (N=3) | Day 1 - Prasugrel (60mg) - Post Infusion (2.0 hr) (N=3) | Day 8 - Prasugrel (10mg) Dosing (6 Doses) (N=6) | Day 8 - Prasugrel (10mg) Dosing (5 Doses) (N=6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site hemmorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — General disorders and administrations site conditions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication or presentation, the Institution will provide the Sponsor thirty (30) days for review and comment, If necessary, Sponsor will be given an additional sixty (60) days to allow Sponsor to file a patent application or taking such other measures as Sponsor deems appropriate to establish and preserve its proprietary rights upon the manuscript or other material for such publication. Sponsor may remove confidential or proprietary information.